CLINICAL TRIAL: NCT02064062
Title: Autologous Stem Cells in Achilles Tendinopathy
Acronym: ASCAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/0419; 2013-000966-12 (EudraCT Number)
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Achilles Tendinitis, Right Leg; Achilles Tendinitis; Achilles Degeneration; Achilles Tendon Thickening; Tendinopathy; Achilles Tendinitis, Left Leg
Keywords: Achilles Tendinopathy; Autologous Stem Cells; Musculoskeletal
MeSH Terms: conditions — Tendinopathy | interventions — SLC25A33 protein, human; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Mesenchymal Stem Cells (Experimental)
  Interventions: Biological: Autologous Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells
  Other Names: Mesenchymal Stem Cells; Stromal Cells; Stem Cells; Cell Therapy

SUMMARY:
This study is looking at a new treatment, using the patient's own stem cells (the repair cells of the body), to see whether this can help reduce pain and promote healing of the Achilles tendon, without side effects.

DETAILED DESCRIPTION:
Tendon disorders compromise pain free activity and often progress to chronic pain with a major impact on quality of life. More than 85,000 patients each year see their general practitioner (GP) with Achilles Tendinopathy (AT) which affects the lower leg in young and middle aged adults. The main treatment is physiotherapy, although surgery is eventually considered in 25-45%of patients, an intervention that requires several months of immobilisation and has unpredictable outcomes.

Other treatments include, shockwave therapy, Platelet Rich Plasma (PRP) (a blood injection of platelet rich plasma) and steroid injections, but other than physiotherapy non have been shown to be better than placebo. There is a need for improved nonsurgical treatments. There is an established treatment in horses that involves injection of the horses own stem cells into the tendon, which has been shown to be effective but has never been used in man. We wish to translate the technology to humans and propose a pilot phase II trial to establish the safety of stem cells implanted in diseased human tendon. We aim to study 10 patients with chronic mid substance achilles tendinopathy to assess safety as our primary outcome measure. In addition we capture clinical outcomes scores and ultrasound appearances. Other than the stem cell injection, all assessments will be non invasive. Participants will be otherwise healthy adults, aged 18-70 and recruited from routine outpatient clinics at the Royal National Orthopaedic Hospital, presenting with a painful heel, diagnosed by a specialist as Achilles tendinopathy, and having already undergone a minimum of 6 months of physiotherapy. Each participant will have 6 months follow up. This study will help inform a larger clinical trial in the future for which a further ethics application will be made.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤ 70 (both males and females)
* Participants with chronic midportion AT (as defined by pain in region of AT and tender swelling in mid portion of AT (no tenderness over bony attachment to heel) with symptoms for longer than 6 months who have failed conservative treatment (at least a full course of physiotherapy) and for whom surgery is being considered
* Able to provide written informed consent

Exclusion Criteria:

* Previous bony surgery (e.g. reconstructive pelvic osteotomy) at or in proximity to the bone marrow harvest site
* Pregnancy or lactation
* Current use of steroids, anti-tumour necrosis factor (TNF) drugs, methotrexate, or ciprofloxacin (or use within 4 weeks of assessment for eligibility)
* Positive for hepatitis B virus (HBV), Hepatitis C virus (HCV), Human Immunodeficiency Virus (HIV 1 and 2), syphilis and human t-cell leukaemia virus (HTLV)
* Previous AT surgery on the tendon to receive mesenchymal stem cell (MSC) implantation
* Inflammatory arthritis
* Known or suspected underlying haematological malignancy
* Other active malignancy in the past 3 years
* Bovine or antibiotic allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The primary safety outcome will be the incidence rate of Serious Adverse Reaction (SAR). | 6 months
  The primary safety outcome is the incidence rate of SARs. This will be expressed as the proportion of participants experiencing a SAR at any time over the 24 week follow-up period. Primary outcomes will be assessed by adverse events reporting, clinical assessment and ultrasound.

SECONDARY OUTCOMES:
Incidence of success | 6 months
  The secondary efficacy outcome measure is the incidence of success at 6 months, where success is defined as a reduction of 2 or more points on VAS of pain and an increase of VISA-A score greater than the Minimum Clinically Important Difference (MCID).
Conventional ultrasound changes from baseline | Baseline immediately before implantation and at weeks 6, 12 and 24
Ultrasound Tissue Characterisation (UTC) changes from baseline | Baseline immediately before implantation and at weeks 6, 12 and 24
Inter-observer reliability of UTC against conventional US | Baseline immediately before implantation and at weeks 6, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Goldberg, MBBS MD FRCSI FRCS(Tr&Orth), Principal Investigator — Royal National Orthopaedic Hospital NHS Trust, UCL
Locations (1):
- Royal National Orthopaedic Hospital, London, United Kingdom

REFERENCES:
- [Background] Smith RK, Korda M, Blunn GW, Goodship AE. Isolation and implantation of autologous equine mesenchymal stem cells from bone marrow into the superficial digital flexor tendon as a potential novel treatment. Equine Vet J. 2003 Jan;35(1):99-102. doi: 10.2746/042516403775467388. No abstract available. PMID 12553472
- [Derived] Goldberg AJ, Zaidi R, Brooking D, Kim L, Korda M, Masci L, Green R, O'Donnell P, Smith R. Autologous Stem Cells in Achilles Tendinopathy (ASCAT): protocol for a phase IIA, single-centre, proof-of-concept study. BMJ Open. 2018 May 14;8(5):e021600. doi: 10.1136/bmjopen-2018-021600. PMID 29764889
- See also: Related Info — http://www.ucl.ac.uk/jro/academic-clinical-trials/advanced-therapies